CLINICAL TRIAL: NCT04058015
Title: Admission Hyperglycemia in Patients With Moderate to Severe Thoracoabdominal Injuries is Associated With Higher Mortality Rate Than Non-Diabetic Normoglycemic Patients
Brief Title: Outcome of Patients With Thoraco-abdominal Injury and Stress-induced Hyperglycemia or Diabetic Hyperglycemia
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201900726B0
Record Dates: First submitted 2019-08-13; First posted 2019-08-15 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-06

CONDITIONS: Abdominal Injury; Thoracic Injury; Hyperglycemia; Hyperglycemia Stress
Keywords: admission hyperglycemia; stress-induced hyperglycemia; diabetic hyperglycemia; diabetes mellitus; thoracoabdominal trauma; mortality
MeSH Terms: conditions — Abdominal Injuries; Thoracic Injuries; Hyperglycemia; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- adult patients with thoracoabdominal injuries: adult patients with moderate to severe thoracoabdominal injuries
  Interventions: Other: Stress-induced hyperglycemia; Other: Diabetic hyperglycemia; Other: Diabetic normoglycemia; Other: Non-diabetic normoglycemia

INTERVENTIONS:
Other: Stress-induced hyperglycemia — Stress-induced hyperglycemia (SIH)was defined as a serum glucose ≥ 200 mg/dL in the patients without Diabetes mellitus.
Other: Diabetic hyperglycemia — Diabetic hyperglycemia (DH) which indicated a serum glucose ≥ 200 mg/dL in patients with Diabetes mellitus.
Other: Diabetic normoglycemia — Diabetic normoglycemia (DN), which was defined when there was a serum glucose < 200 mg/dL in the patients with Diabetes mellitus.
Other: Non-diabetic normoglycemia — Non-diabetic normoglycemia (NDN) indicating a serum glucose < 200 mg/dL in patients who were absent of Diabetes mellitus.

SUMMARY:
This study aimed to measure the effects of SIH and DH on the mortality outcomes of the adult patients with moderate to severe thoracoabdominal injury

DETAILED DESCRIPTION:
Because the pathophysiologic response of the patients with a thoracoabdominal injury is different from those who had a traumatic brain injury, this study aimed to measure the effects of hyperglycemia induced by stress or by diabetes on the outcomes of patients with thoracoabdominal injuries in comparison with those who had non-diabetic normoglycemia (NDN). The primary study hypothesis stated that, following thoracoabdominal injuries, the patients with SIH had a worse outcome than patients with DH. The primary outcome was mortality rate of these patients.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with moderate to severe thoracoabdominal injuries

Exclusion Criteria:

* patients with a thoracic and abdominal abbreviated injury scale (AIS) < 3
* patients who had polytrauma which was defined as there was additional AIS scores ≥ 3 points in other regions of the body
* patients less than 20 years old
* patients who had sustained a burn injury

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective study reviewed data from trauma patients registered between January 1, 2009 and December 31, 2018. The inclusion criteria were age ≥20 years Adult patients with moderate to severe thoracoabdominal injuries (n = 802) were grouped into four exclusive subgroups: (1) SIH, which was defined as a serum glucose ≥ 200 mg/dL in the patients without DM (n = 52); (2) DH, which indicated a serum glucose ≥ 200 mg/dL in patients with DM (n = 79); (3), DN, which was defined when there was a serum glucose < 200 mg/dL in the patients with DM (n = 50); and (4) NDN, indicating a serum glucose < 200 mg/dL in patients who were absent of DM (n = 621)
Sampling Method: Probability Sample
Enrollment: 802 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-08-09 (Actual)

PRIMARY OUTCOMES:
in-hospital mortality | up to 6 months
  The primary outcome of the study was in-hospital mortality.

CONTACTS AND LOCATIONS:
Overall Officials: TSANG-TANG Hsieh, Study Chair — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan